CLINICAL TRIAL: NCT02565927
Title: A Novel Tracheal Radioactive Stent Loaded With 125I Seeds for the Malignant Airway Obstruction Versus a Conventional Stent: A Prospective Randomized Controlled Trial
Brief Title: A Trail of a Novel Tracheal Radioactive Stent for the Malignant Airway Obstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of Department of Interventional Radiology & Vascular Surgery, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015ZDSYLL032.0
Record Dates: First submitted 2015-09-20; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Malignant Airway Obstruction
Keywords: Trachea; Stent; Intraluminal brachytherapy
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radioactive stent (Experimental): Patients diagnosed as MAO treated with radioactive airway stent loaded with Iodine-125 seeds
  Interventions: Device: Traditional airway stent; Drug: Iodine-125 seeds
- Traditional airway stent (Active Comparator): Patients diagnosed as MAO treated with traditional airway stent
  Interventions: Device: Traditional airway stent

INTERVENTIONS:
Device: Traditional airway stent — process airway stenting
  Other Names: Tracheal stent(Nanjing MicroInvasive Medical Inc.)
Drug: Iodine-125 seeds — process intraluminal brachytherapy
  Other Names: Radioactive seeds(Chinese Atomic Energy Science Institution)
  Arms: Radioactive stent

SUMMARY:
The aim of this study was to evaluate the safety and effectiveness of an radioactive airway stent loaded with 125I seeds compared to a conventional airway stent in patients with malignant airway obstruction caused by both primary and metastatic malignant tumors.

DETAILED DESCRIPTION:
Malignant tumors of the lung, esophagus, thyroid, or other mediastinal structures often involve the trachea by direct tumor growth compression and (or) invasion. In addition, extrathoracic cancers metastasize to these lymph nodes as well. However, surgical resection and airway reconstruction are the gold-standard treatment for MAO, many patients with airway involvement are poor surgical candidates based on physiologic or oncologic criteria.There are three main types of malignant airway obstruction: endobronchial obstruction, extrinsic compression, and a mixed pattern. For endobronchial obstruction, ablative techniques that destroy tissue are indicated, including lasers, electrocautery, argon plasma coagulation (APC), photodynamic therapy, microdebriders, and cryotherapy, but primary tracheal cancers are less common than other types of lung cancer. If the obstruction is exclusively or mainly due to compression from outside the airway wall, the only option consists of placement of a stent or endoprosthesis. However, follow-up data has demonstrated that postoperative restenosis of stenting occurs in 5-45% of cases as a result of neoplastic infiltration through the mesh into the lumen or tumor overgrowth above and below the mesh stents. Encouraged by the success of 125I esophageal and biliary stent in esophageal carcinoma , a tracheal stent loaded with 125I radioactive seeds was developed in investigators'institute. After successful in vitro and in vivo evaluations of the delivery system, investigator will prospectively compare responses to treatment with this irradiation tracheal stent versus the conventional self-expandable stent in patients with MAO.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 80 years
2. MAO caused by any adenocarcinoma with histologically or cytologically confirmation by biopsy or previous surgical procedures
3. symptoms such as dyspnea related to biliary obstruction
4. unresectability or refusal to be surgically treated
5. willing and able to comply with the study procedures and provide written informed consent to participate

Exclusion Criteria:

1. patients with suspected benign airway obstruction
2. airway obstruction that could not be dilated enough to pass the delivery system
3. perforation of any ducts within the tracheal tree
4. presence of metallic tracheal stent or airway surgery
5. acute or chronic inflammation in the airway
6. uncooperative or could not provide authorization and signature.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
diameter stenosis | Participants will be followed till die or lost to follow-up,an expected average of a year.
  reference tracheal diameter minus minimum diameter at stenosis site / reference tracheal diameter×100

SECONDARY OUTCOMES:
Over survival | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Time from stenting to the day when the patients died or lost to the follow-up.

OTHER OUTCOMES:
Success rate | Participants will be followed till die or lost to follow-up,an expected average of a year.
  The rate of relief of the symptoms and signs of the patients
Number of participants with abnormal laboratory values that are telated to treatment | Participants will be followed till die or lost to follow-up,an expected average of a year.
  laboratory examination of white blood cells, IgA, IgG and IgM.
Number of participants with adverse events that are telated to treatment | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Adverse events as follows: severe chest pain, hemoptysis, perforation, pneumonia
dyspnea index | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Dyspnea index grades are as follows: grade 0,asymptomatic while climbing stairs; grade I, symptomatic climbing stairs; grade II, symptomatic after walking 100 m on flat ground; grade III, symptomatic with the least effort (talking,getting dressed); and grade IV, symptomatic in bed, at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China